CLINICAL TRIAL: NCT01796366
Title: A Multiple Dose Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC0123-0000-0338 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1953-4013; 2012-003046-32 (EudraCT Number); U1111-1132-0943 (Other: WHO)
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin 338 + placebo (Experimental)
  Interventions: Drug: insulin 338 (GIPET I); Drug: placebo
- Insulin glargine + placebo (Active Comparator)
  Interventions: Drug: insulin glargine; Drug: placebo

INTERVENTIONS:
Drug: insulin 338 (GIPET I) — Each subject will be allocated to one of three dosing periods only. The subject will receive oral insulin 338 and placebo, administered subcutaneously (s.c., under the skin) once daily for 10 days at fixed dose levels.
  Arms: Insulin 338 + placebo
Drug: placebo — S.c placebo administered in combination with insulin 338
  Arms: Insulin 338 + placebo
Drug: insulin glargine — Each subject will be allocated to one of three dosing periods only. The subject will receive insulin glargine for s.c. administration and oral placebo once daily for 10 days at fixed dose levels.
  Arms: Insulin glargine + placebo
Drug: placebo — Oral placebo administered in combination with s.c. insulin glargine
  Arms: Insulin glargine + placebo

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of NNC0123-0000-0338 (insulin 338) in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male subject, or female subject of no childbearing potential, if surgically sterilized (i.e. tubal ligation, bilateral oopherectomies (removal of both ovaries and both fallopian tubes) or hysterectomised) for at least 3 months or if postmenopausal (i.e. as defined by amenorrhoea for at least 12 months prior to screening and documented by follicle stimulating hormone (FSH) levels above 40 U/L)
* Body mass index (BMI) between 20.0 and 35.0 kg/m^2 (both inclusive)
* Type 2 diabetes mellitus (as diagnosed clinically) for 12 months or more

Exclusion Criteria:

* Known or suspected hypersensitivity to trial products or related products
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea) within 2 weeks prior to dosing, as judged by the Investigator
* Any chronic disorder or severe disease which in the opinion of the Investigator might jeopardise subject's safety or compliance with the protocol

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2013-08-19 (Actual); Study Completion 2013-08-19 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | As recorded from first trial product administration (Day 1) and until Sub-visit 2A (Day 12) of the dosing visit

SECONDARY OUTCOMES:
Area under the serum insulin concentration-time curve | During one dosing interval (0-24 hours) at steady-state (Day 10)
Area under the glucose infusion rate-time curve | During one dosing interval (0-24 hours) at steady state (Day 10)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com